CLINICAL TRIAL: NCT03373071
Title: Phase I/II Study of Anti-CD19 Chimeric Antigen Receptor-Expressing T Cells in Pediatric Patients Affected by Relapsed/Refractory CD19+ Acute Lymphoblastic Leukemia and Non Hodgkin Lymphoma
Brief Title: Anti-CD19 CAR T Cells in Pediatric Patients Affected by Relapsed/Refractory CD19+ ALL and NHL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Franco Locatelli, Haematology-Oncology Department Chief, Bambino Gesù Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-CAR01
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: CD19-ALL; CD19-LNH
Keywords: CD19-CAR T cell; CD19-malignancy; CAR T cell; CD19-ALL; CD19-LNH

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19-CART01 (Experimental): Following the lymphodepleting treatment, with patients will be treated with 0.5 to 3.0 x 10⁶/kg CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose
  Interventions: Biological: CD19-CAR T cell

INTERVENTIONS:
Biological: CD19-CAR T cell — Following lymphodepletion with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with 0.5 to 3.0 x 10⁶/kg CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.
  In case of toxicity, the patient will receive the dimerizing drug activating the suicide safety switch in order to improve the safety of the treatment

SUMMARY:
The primary objective of this phase I study is to evaluate the safety and to establish the recommended dose of CD19-CART01 infused in pediatric patients affected by relapsed/refractory B-ALL or NHL with measurable Bone Marrow (BM) involvement. The phase II extension is aimed at testing the efficacy of the treatment at the optimal dose defined in the phase I.

DETAILED DESCRIPTION:
The study will consist of 2 phases, a Phase I or dose escalation phase and a Phase II or expansion phase. Paediatric/young adult patients with relapsed or refractory B cell ALL will be enrolled. Eligible patients will undergo leukapheresis in order to harvest T cells, which is the starting material for the manufacture. Autologous CAR T product directed against CD19-expressing tumor cells (CD19-CART01) will be produced and, after a lymphodepletion with conventional chemoterapic agents, the patient will receive CD19-CART01 intravenously. The construct contains also the suicide gene safety switch "inducible Caspase 9"; therefore, in case of relevant toxicities, the patient will receive the dimerizing agent in order to induce the apoptosis of the cells.

After the treatment, the patients will then enter a 36-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with CD19 expressing B-cell acute lymphoblastic leukemia (ALL) or Non-Hodgkin Lymphoma (NHL) with BM involvement and one of the following:

   i. Patients in 2nd or subsequent relapse, after at least one standard frontline chemotherapy and one salvage regimen, with BM involvement ii. Relapse after allogeneic HSCT, if at least 100 days post-transplant, if there is no evidence of active GVHD and if the patient is no longer taking immunosuppressive agents for at least 30 days prior to enrollment iii. MRD > 0.1% after either reinduction therapy or any course of consolidation for relapsed ALL
2. Measurable or evaluable disease at the time of enrollment, which may include any evidence of disease, including MRD detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
3. Age: 6 months - 25 years.
4. Voluntary informed consent is given. For subjects < 18 year-old their legal guardian must give informed consent. Pediatric subjects will be included in age-appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate.
5. Clinical performance status: Patients > 16 years of age: Karnofsky greater than or equal to 60%; Patients < 16 years of age: Lansky scale greater than or equal to 60%.
6. Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
7. Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.

Exclusion Criteria:

1. Pregnant or lactating women
2. Severe, uncontrolled active intercurrent infections
3. HIV, or active HCV and/or HBV infection
4. Life-expectancy < 6 weeks
5. Hepatic function: Inadequate liver function defined as total bilirubin > 4x upper limit of normal (ULN) or transaminase (ALT and AST) > 6 x ULN
6. Renal function: serum creatinine > 3x ULN for age.
7. Blood oxygen saturation < 90%.
8. Cardiac function: Left ventricular ejection fraction lower than 45% by ECHO.
9. Congestive heart failure, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject.
10. BM blasts > 50% pre-infusion.
11. Hyperleukocytosis (greater than or equal to 20,000 blasts/microliter) or rapidly progressive disease that in the evaluation of the investigator would compromise ability to complete study therapy
12. Active CNS disease as documented by the presence of blasts in the CSF or by MRI. This criterion could be revised once that, after the phase I portion of the study, absence of life-threatening (i.e. grade IV) neurological toxicity will be documented.
13. Presence of active, grade 2-4 acute or extensive chronic GvHD
14. Recurrent or refractory ALL with testicular involvement
15. Concurrent or recent prior therapies, before infusion:

    i. Systemic steroids (at a dose > 2 mg/kg prednisone) in the 2 weeks before infusion. Recent or current use of inhaled/topical/non-absorbable steroids is not exclusionary.

    ii. Systemic chemotherapy in the 2 weeks preceding infusion. iii. Anti-thymocyte globulin (ATG) or Alemtuzumab (Campath®) in the 4 weeks preceding infusion.

    iv. Immunosuppressive agents in the 2 weeks preceding infusion. v. Radiation therapy must have been completed at least 3 weeks prior to enrollment.

    vi. Other anti-neoplastic investigational agents currently administered or within 30 days prior to infusion (i.e. start of protocol therapy);

    vii. Exceptions:
    1. There is no time restriction with respect to prior intrathecal chemotherapy, provided that there is complete recovery from any acute toxic effects of such;
    2. Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study provided that they meet all other eligibility criteria;
    3. Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided that there has been no increase in dose for at least 2 weeks prior to starting apheresis;
16. Patient-derived CD19-CART01 production failure

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-23 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Phase I - Identification of the dose limiting toxicity (DLT) | 4 weeks after CAR T cell infusion
  Toxicity will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) scale, version 4 and the number of patients experiencing DLT will be evaluated
Phase II - Efficacy | 4 weeks after CAR T cell infusion
  Complete remission rate minimal residual disease (MRD) negative response

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 4 weeks after CAR T cell infusion
  Assessment of CR with incomplete blood count recovery (CRi), Partial Response (PR) and Stable Disease (SD).
In vivo persistence/expansion of infused CAR T cell | Up to 5 years
  Detection of infused CAR T cell in the peripheral and bone marrow blood
Function of infused CAR T cell | Up to 5 years
  Assessment through functional assays (such as ELISPOT for interferon-gamma release using CD19-positive cells and CD19-negative target cells) and immunophenotyping on peripheral blood mononuclear cells (PBMCs) isolated from the patients
Cytokine profiling | 10 days after CAR T cell infusion
  Define serum cytokine profile after T cell infusion and correlation with cytokine release syndrome (CRS)
Disease Outcome | Up to 3 years
  Assessment of relapse rate
Overall Survival | Up to 3 years
Disease-free survival | Up to 3 years
Elimination of CAR T cell in case of toxicity | Up to 15 years
  Assessment the kinetics of CAR T cells elimination after AP1903 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338